CLINICAL TRIAL: NCT02956694
Title: Design, Implementation and Evaluation of a Tailored Intervention to Improve Shared Decision Making Among Seniors With Dementia, Their Caregivers and Healthcare Providers
Brief Title: Intervention to Improve Shared Decision Making Among Seniors With Dementia, Their Caregivers and Healthcare Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anik Giguère (Other)
Collaborators: Ministère de l'Économie, de l'Innovation et de l'Exportation du Québec (Unknown); SOVAR (Unknown); Laval University (Other)
Responsible Party: Sponsor-Investigator, Anik Giguère, Assitant Professor, Laval University
Organization: Laval University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-2015-PSVT2-31404
Record Dates: First submitted 2016-10-31; First posted 2016-11-07 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Dementia; Professional-Patient Relations; Professional-Family Relations; Aging
Keywords: Aged; Cognitive impairment; Neurocognitive Disorders; Shared decision making; Distance learning; Primary care; Decision support tool; Patient decision aid
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: We evaluated the effectiveness of the intervention, here a training program, using a pre-post design, and also assessed the barriers and facilitators to completing the training program.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Professional training (Experimental): Professional e-learning program on shared decision making including two components: (1) a self-directed e-learning activity on shared decision making, lasting about 1 hour, that participants could complete in several sittings; and (2) five evidence summaries named Decision Boxes (DBs).
  Interventions: Behavioral: Professional e-learning program on shared decision making

INTERVENTIONS:
Behavioral: Professional e-learning program on shared decision making — Clinicians will have access to a, e-learning program on shared decision making (e-TUDE) during one month. They will also receive five Decision Boxes (DB) dealing with difficult decisions often faced by seniors with dementia and their caregivers in primary care. They will receive five DBs by email, at a rate of 1 per week for 5 weeks.

SUMMARY:
The increasing prevalence of Alzheimer's disease and other forms of dementia causes new challenges to ensure that healthcare decisions are informed by research evidence and reflect what is important for seniors and their caregivers. Primary care providers point to a need for more training on communication with families of seniors living with dementia, and on the non-pharmacological health options that are often recommended before use of medications.Therefore, the investigators will design and evaluate an intervention to train primary healthcare providers on how to empower seniors with dementia and their caregivers in making health-related decisions based on research evidence and on their preferences and priorities. A distance professional training program on shared decision making will initially be designed, comprising evidence summaries to be shared with patients living with dementia and their caregivers who face difficult decisions. Patients with dementia, their caregivers and healthcare providers, will then provide feedback on the training program, which will then be improved following their suggestions. In a last step, the investigators will study the processes required to implement this training program and measure its effects on provider knowledge and intention to adopt shared decision making.

DETAILED DESCRIPTION:
Background: The increasing prevalence of Alzheimer's disease and other forms of dementia causes new challenges in primary care. Indeed, primary care providers point to a need for more training to care for this population, especially seniors presenting behavioural and psychological symptoms of dementia. They also find the inter-professional nature of care, and the need to communicate with community services and families, very challenging. Moreover, patients living with dementia and their caregivers consistently report their need for more information about dementia. Therefore, in a recent survey, the investigators sought five difficult decisions that patients living with dementia and their informal caregivers often face in primary care settings. In the current study, they propose to tailor and evaluate an e-learning professional training program on shared decision making, comprising evidence summaries on the health options to consider before making these five difficult decisions. This tailored training program is expected to improve shared decision making between clinicians and patients with dementia and their caregivers, and in turn improve patient and caregiver empowerment in relation to their own health care.

Methods: In two phases, the aims of this study are to (1) design and tailor the intervention, and (2) implement and evaluate it. In the first phase, theory and user-centred design will be used to tailor a multifaceted intervention comprising a distance professional training program on shared decision making, and five shared decision-making tools dealing with difficult decisions often faced by seniors with dementia and their caregivers. Each tool will be designed in two versions, one for clinicians, and one for patients/caregivers. Forty-nine clinicians and 27 patients/caregivers will be invited to participate to three cycles of design-evaluation-feedback of each intervention components. Besides think-aloud and interview approaches, they will also complete questionnaires to identify the factors most likely to influence their adoption of shared decision making after exposure to the intervention. Thereafter, the intervention will be modified by adding/enhancing behaviour-change techniques targeting these factors. In the second phase, the effectiveness of this tailored intervention will be evaluated before/after implementation, in a two-armed, clustered randomized trial with a three-month follow-up. A convenience sample of primary care clinics and home care services will be enrolled in the province of Quebec (Canada), and health care providers who practice there will be recruited (mostly family physicians, nurses, and social workers). We will record participants' access to training component, and conduct telephone interviews with a purposeful sample of participants, half of whom completed training and the other half whom did not. The participants will also complete a survey before and after training, to assess their knowledge, and intention to adopt shared decision making. Three researchers will conduct a thematic qualitative analysis of the interviews, as per the theory of planned behaviour. We performed bivariate analyses with the survey data.

Discussion: The results of this study will allow modifying the training program to improve participation rates and, ultimately, uptake of meaningful sjared decision making with patients living with dementia.

ELIGIBILITY:
Inclusion criteria:

Healthcare professionals from various professions (e.g., family physicians, nurses, and social workers) who practice in family medicine clinics and homecare services in the province of Quebec, Canada.

Exclusion criteria:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Change in healthcare providers' intention to adopt shared decision making | Right before training, and then one week after the end of training
  Participants' intention to use shared decision making with their next patient facing a preference-sensitive decision, and the determinants of this intention (attitude, beliefs about capabilities, moral norm, and social influence), using a brief 5-item version of the CPD-REACTION (Légaré et al. Development of a Simple 12-Item Theory-Based Instrument to Assess the Impact of Continuing Professional Development on Clinical Behavioral Intentions. PLoS One. 2014; 9(3): e91013.
Change in healthcare providers' knowledge | Right before training, and then one week after the end of training
  This outcome comprises: knowledge about shared decision making, knowledge about risk communication, perceived awareness of the options. It also comprises variables to assess clinical knowledge on deprescribing anti-psychotics, on the impacts of stopping driving, on the strategies to communicate about stopping driving, on the risk factors for caregiver burden, on the awareness of the information to provide patients to reflect upon the power of attorney, on the elements to check prior to recommending a treatment to a vulnerable senior.
  Two questions were inspired by the Ottawa Decision Support Framework to assess participants' knowledge about SDM (https://decisionaid.ohri.ca/docs/develop/ODSF.pdf); and 10 questions included case-based scenarios,to assess clinical knowledge relative to the care of older adults living with NCD, and reflected the basic principles to develop constructed-response items [28].
Change in Healthcare providers' role preference | Right before training, and then one week after the end of training
  Healthcare professionals' preferred role in decision-making (Strull WM, Lo B, Charles G. Do patients want to participate in medical decision making? JAMA.

CONTACTS AND LOCATIONS:
Overall Officials: Anik MC Giguere, PhD, Principal Investigator — Laval University
Locations (1):
- Réseau de Recherche Axée sur les Pratiques de Première Ligne Université Laval (RRAPPL-UL), Québec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after the study is published.
Access Criteria: Contact the trial sponsor at anik.giguere@fmed.ulaval.ca

REFERENCES:
- [Derived] Giguere AMC, Lawani MA, Fortier-Brochu E, Carmichael PH, Legare F, Kroger E, Witteman HO, Voyer P, Caron D, Rodriguez C. Tailoring and evaluating an intervention to improve shared decision-making among seniors with dementia, their caregivers, and healthcare providers: study protocol for a randomized controlled trial. Trials. 2018 Jun 25;19(1):332. doi: 10.1186/s13063-018-2697-1. PMID 29941020